CLINICAL TRIAL: NCT06793189
Title: A Prospective Study to Evaluate the Efficacy and Safety of MZL-IPI Risk-adapted Targeted Therapy in Patients With Untreated Marginal Zone B-cell Lymphoma
Brief Title: MZL-IPI Risk-adapted Targeted Therapy in Untreated MZL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor and Director，Shanghai Institute of Hematology, Ruijin Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAGIC
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Marginal Zone Lymphoma(MZL)
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — obinutuzumab; orelabrutinib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obinutuzumab and Orelabrutinib (O2) regimen (Experimental): Low-risk patients (MZL-IPI 0-2 points)
  Interventions: Drug: Obinutuzumab and Orelabrutinib; Drug: Orelabrutinib
- Obinutuzumab, Orelabrutinib and Lenalidomide (O2R) regimen (Experimental): High-risk patients (MZL-IPI 3-5 points)
  Interventions: Drug: Obinutuzumab, Orelabrutinib and Lenalidomide; Drug: Orelabrutinib

INTERVENTIONS:
Drug: Obinutuzumab and Orelabrutinib — Induction: Obinutuzumab (1000 mg on days 1, 8, and 15 of cycle 1; 1000 mg on day 1 of cycles 2-6, cycle length=21 days) and Orelabrutinib (150 mg once daily).
  Arms: Obinutuzumab and Orelabrutinib (O2) regimen
Drug: Obinutuzumab, Orelabrutinib and Lenalidomide — Induction: Obinutuzumab (1000 mg on days 1, 8, and 15 of cycle 1; 1000 mg on day 1 of cycles 2-6, cycle length=21 days), Orelabrutinib (150 mg once daily), and Lenalidomide (25 mg on days 2-11 of cycles 1-6, cycle length=21 days).
  Arms: Obinutuzumab, Orelabrutinib and Lenalidomide (O2R) regimen
Drug: Orelabrutinib — Maintenance: Orelabrutinib monotherapy (150 mg once daily up to 24 months).
  Arms: Obinutuzumab and Orelabrutinib (O2) regimen
Drug: Orelabrutinib — Maintenance: Orelabrutinib monotherapy (150 mg once daily up to 24 months).
  Arms: Obinutuzumab, Orelabrutinib and Lenalidomide (O2R) regimen

SUMMARY:
Marginal zone lymphoma (MZL) is a common type of indolent lymphoma that originates from the marginal zone of lymphoid follicles. This study aims to evaluate targeted therapy based on the prognostic risk stratification of MZL-IPI in newly diagnosed MZL cases requiring systemic treatment, and provides a basis for precision treatment of MZL.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histopathologically confirmed CD20-positive marginal zone lymphoma (according to the 2016 WHO classification).

  2. Age ≥ 18 years old, regardless of gender. 3. MZL patients requiring systemic treatment, including but not limited to:
  1. Helicobacter pylori (HP)-positive or HP - negative gastric mucosa extranodal marginal zone lymphoma (MALT) patients with progression/relapse after local treatment (including surgery, radiotherapy, and anti - Helicobacter pylori treatment).
  2. Non - gastric MALT patients with Ann Arbor stage I - II who have progression/relapse after local treatment (including surgery, radiotherapy, etc.), or untreated patients with Ann Arbor stage III - IV who meet the GELF criteria recommended by the NCCN guidelines.
  3. Splenic marginal zone lymphoma (SMZL) patients with progression/relapse after local treatment (including splenectomy, antiviral treatment for HCV - positive patients, etc.), or untreated patients meeting the criteria of progressive or painful splenomegaly, symptomatic or progressive cytopenia such as HB < 100g/L, PLT < 80×10⁹/L, absolute neutrophil count (ANC) < 1.0×10⁹/L.
  4. Nodal marginal zone lymphoma (NMZL) patients with Ann Arbor stage I - II who have progression/relapse after local treatment (including surgery, radiotherapy, etc.), or untreated patients with Ann Arbor stage III - IV who meet the GELF criteria recommended by the NCCN guidelines.

  4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2. 5. Life expectancy of at least 3 months. 6. The patient has adequate bone marrow (except those caused by MZL), liver and kidney functions.

  7. Able to comply with the research procedures and cooperate in the implementation of the entire research process; 8. Written informed consent; 9. Women with fertility agree to take appropriate measures to avoid pregnancy during the treatment period until at least one year after the end of treatment; Men agree to maintain abstinence or use barrier contraception.

Exclusion Criteria:

* 1. Histologically transformed into high-grade lymphoma. 2. Known central nervous system involvement of MZL. 3. Previous systemic treatment including immunotherapy, chemotherapy or targeted drugs.

  4. Previous autologous stem-cell transplantation or allogeneic tissue/solid organ transplantation.

  5. History of other invasive cancers within the past 3 years that have not received curative treatment or are still receiving anti-cancer treatment (including hormonal therapy for breast or prostate cancer).

  6. Complicated with uncontrolled cardiovascular and cerebrovascular diseases (such as New York Heart Association-defined grade 3 or 4 heart failure, arrhythmia, myocardial infarction, stroke, or intracranial hemorrhage), coagulation - disorder diseases, connective tissue diseases, severe infectious diseases (including active pulmonary tuberculosis), etc.

  7. Known human immunodeficiency virus (HIV) infection, or active hepatitis B or C virus infection (positive result shown by polymerase chain reaction [PCR]). Serological antibody - positive is allowed if HBV DNA < 10³ IU/ml; HCV RNA test must be negative.

  8. Vaccinated with live attenuated vaccines within 4 weeks before starting investigational treatment. During the study, patients are prohibited from receiving live attenuated vaccine inoculations, including influenza vaccines.

  9. Requiring continuous treatment with potent and moderate-effect CYP3A inhibitors or CYP3A inducers.

  10. Unable to swallow capsules or having diseases that significantly affect gastrointestinal function, such as malabsorption syndrome, bariatric surgery, inflammatory bowel disease, or partial or complete intestinal obstruction.

  11. Psychiatric patients or other patients known or suspected to be unable to fully comply with the study protocol.

  12. Pregnant or lactating women. 13. Other concurrent and uncontrolled medical conditions that, in the investigator's opinion, will affect the patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2025-01-21 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival | Baseline up to data cut-off (up to 24 months).
  Progression-free survival is defined as the time from registration to the first occurrence of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first; as assessed by the investigator.

SECONDARY OUTCOMES:
Complete Response Rate after 6 cycles, at 12 months and 24 months | At the end of cycle 6, at 12 months and 24 months after treatment start.
  The proportion of patients with complete response after 6 cycles, 12 months and 24 months from treatment start, according to the 2014 Lugano Response Criteria.
Overall Response Rate after 6 cycles, at 12 months and 24 months | At the end of cycle 6, at 12 months and 24 months after treatment start.
  The proportion of patients with complete and partial response after 6 cycles, 12 months and 24 months from treatment start, according to the 2014 Lugano Response Criteria.
Treatment-Related Adverse Events rate as assessed by CTCAE version 5.0 | From enrollment to study completion (up to approximately 24 months).
Duration of Response (DOR) | From enrollment to study completion (up to approximately 24 months).
  Duration of response is defined as the period from the first response (at least PR) to treatment until evidence of disease progression, relapse or death of any cause.
Histological transformation rate | From enrollment to study completion (up to approximately 24 months).
  Histological transformation rate is defined as the proportion of patients with histological transformation.
2-year overall survival | Baseline up to data cut-off (up to 24 months).
  Overall survival is defined as the time from registration to death from any cause.